CLINICAL TRIAL: NCT01566318
Title: Depression Agency-Based Collaborative (Depression ABC)
Brief Title: Depression Agency-Based Collaboration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Steven M. Albert, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P30MH090333-PRC1; P30MH090333 (NIH)
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Major Depression; Anxiety Disorder
Keywords: Depression; Anxiety; Geriatric mental health
MeSH Terms: conditions — Depressive Disorder, Major; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Problem solving therapy (PST) (Experimental): 6-8 sessions of PST, with booster, delivered over 8 weeks
  Interventions: Behavioral: Problem-Solving Therapy
- Usual care (No Intervention): Usual agency care, monitored for mental health services

INTERVENTIONS:
Behavioral: Problem-Solving Therapy — 6-8 sessions over 8 weeks, with booster
  Arms: Problem solving therapy (PST)

SUMMARY:
Seniors who receive supportive services face a variety of psychosocial vulnerabilities that put them at risk for depression. One group with very high risk is older adults receiving aging services through Medicaid waiver programs. This 3-year research uses a randomized controlled clinical trial to assess the effectiveness of brief behavioral therapies (problem solving therapy [PST] and Brief Behavioral Therapy for Insomnia [BBTI]) to prevent depression in seniors receiving aging services.

DETAILED DESCRIPTION:
The research will determine (i) if a course of problem solving therapy (PST) and Brief Behavioral Therapy for Insomnia (BBTI), with boosters, reduces incidence of major depressive episodes over 12 months relative to usual care, and (ii) the extent to which behavioral therapies achieve these effects through enhancement of protective factors, such as greater self-efficacy, better targeting of services to address needs, and greater control over home environments.

Periodic blood draws will be used to assess biosignatures of depression. Guiding our investigations of pharmacogenetics, inflammation, and proteomics are synergistic interactions among the serotonergic system, the HPA axis, systemic inflammation, growth factors such as brain derived neuro-trophic factor (BDNF), psychosocial stressors, and vascular co-morbidity. Genetic variation in vasopressin receptors, potentially involved in both cardiovascular risk and social attachment, is also associated with recurrence of depression. Similarly, genetic variation in inflammation may influence antidepressant response and medical co-morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Age => 60 years
* Modified Mini Mental State (3MS) Examination =>80
* Receiving aging services or difficulty with 1+ ADL/IADL
* PHQ-9 score > 0 and <= 9 (and question 1 or 2 is >0)

Exclusion Criteria:

* Major depressive episode or anxiety disorder within 12 mo
* Ever diagnosed with bipolar disorder or schizophrenia
* Drug or alcohol use disorder within the past 12 months
* Currently taking antidepressants
* Currently taking antianxiety med >4x/week for past 4 weeks

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2012-03; Primary Completion 2016-02 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Major depressive disorder | 12 months
  Patient Health Questionnaire score > 9 with confirming diagnostic interview
Generalized anxiety disorder | 12 months
  Generalized anxiety disorder score >=10, and meets criteria for SCID or PRIME-MD diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Albert, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] van't Veer-Tazelaar PJ, van Marwijk HW, van Oppen P, van Hout HP, van der Horst HE, Cuijpers P, Smit F, Beekman AT. Stepped-care prevention of anxiety and depression in late life: a randomized controlled trial. Arch Gen Psychiatry. 2009 Mar;66(3):297-304. doi: 10.1001/archgenpsychiatry.2008.555. PMID 19255379